CLINICAL TRIAL: NCT03612180
Title: Evaluation of Metoprolol Pharmacokinetics in Patients Receiving Hi Flux Hemodialysis
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Amy Barton Pai, Amy Pai PharmD Associate Professor, University of Michigan
Other Study IDs: HUM00138192
Record Dates: First submitted 2018-07-12; First posted 2018-08-02 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Hemodialysis; Pharmacokinetics
MeSH Terms: interventions — Metoprolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Metoprolol Succinate — Pharmacokinetics

SUMMARY:
The current study will evaluate the plasma pharmacokinetics of metoprolol in a cohort of 8 adult volunteers who are receiving regular hemodialysis treatment (HD) 3 days a week for 4 hours each day and have been taking a total daily dose of 25-200 mg of metoprolol succinate for >30 days as part of their usual care. Blood sampling will occur over 10 hours, with frequent sampling during HD and in the 4 hours after termination of HD treatment. The 8 subjects will all receive their prescribed dose (25-200 mg total daily dose) 2 hours prior to HD treatment. The pre-HD sample will also be sent for pharmacogenomics genotyping. Safety and pharmacodynamic assessments (blood pressure (BP) and heart rate (HR) assessments) will be performed throughout the study. Axiom Precision Medicine Research Array (Affymetrix, Santa Clara, CA) will be used to evaluate genotype of CYP2D6. CYP2D6 phenotype will be evaluated using the ratio of parent drug to metabolite. Non-compartmental analyses will be performed to compare maximum concentrations (Cmax), time to maximum concentration and area under the curve from time 0 to the last measurable sample (AUClast) between the two phases. Compartmental analyses will be performed to construct a model to explain time-dependent changes in metoprolol clearance. Monte Carlo simulations will be performed to compare metoprolol pharmacokinetic profiles on and off HD.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Indwelling tunneled catheter, AVF, AVG that is currently used for hemodialysis
3. Receiving in-center hemodialysis 3 days a week for 3-4.5 hours each treatment
4. Taking a total daily dose of 25-200 mg metoprolol succinate as prescribed by their physician
5. Hemoglobin ≥ 9.5 g/dL on most recent laboratory assessment prior to study

Exclusion Criteria:

1. Any condition that would not allow for arm BP to be taken
2. Hemoglobin < 9.5 g/dL on most recent lab prior to study
3. Patient is on a CYP2D6 inhibitor (most common in HD population amiodarone, bupropion, cinacalcet, diphenhydramine, fluoxetine, paroxetine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory in-center hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics-Maximal Plasma Concentration | Pre-dialysis, during dialysis (30 minutes, 2 hours, end of treatment) and post-dialysis (30 minutes, 2 hours and 4 hours)
  Characterize the pharmacokinetics of metoprolol and its metabolite, alpha-hydroxymetoprolol during and after HD
Plasma pharmacokinetics-Time to Maximal Plasma Concentration | Pre-dialysis, during dialysis (30 minutes, 2 hours, end of treatment) and post-dialysis (30 minutes, 2 hours and 4 hours)
  Characterize the pharmacokinetics of metoprolol and its metabolite, alpha-hydroxymetoprolol during and after HD
Plasma Pharmacokinetics-Area under the concentration time curve (AUC) | Pre-dialysis, during dialysis (30 minutes, 2 hours, end of treatment) and post-dialysis (30 minutes, 2 hours and 4 hours)
  Characterize the pharmacokinetics of metoprolol and its metabolite, alpha-hydroxymetoprolol during and after HD
Plasma Pharmacokinetics-Clearance | Pre-dialysis, during dialysis (30 minutes, 2 hours, end of treatment) and post-dialysis (30 minutes, 2 hours and 4 hours)
  Characterize the pharmacokinetics of metoprolol and its metabolite, alpha-hydroxymetoprolol during and after HD
Plasma Pharmacokinetics-Volume of Distribution | Pre-dialysis, during dialysis (30 minutes, 2 hours, end of treatment) and post-dialysis (30 minutes, 2 hours and 4 hours)
  Characterize the pharmacokinetics of metoprolol and its metabolite, alpha-hydroxymetoprolol during and after HD
Plasma Pharmacokinetics-elimination rate constant | Pre-dialysis, during dialysis (30 minutes, 2 hours, end of treatment) and post-dialysis (30 minutes, 2 hours and 4 hours)
  Characterize the pharmacokinetics of metoprolol and its metabolite, alpha-hydroxymetoprolol during and after HD
Plasma Pharmacokinetics-half-life | Pre-dialysis, during dialysis (30 minutes, 2 hours, end of treatment) and post-dialysis (30 minutes, 2 hours and 4 hours)
  Characterize the pharmacokinetics of metoprolol and its metabolite, alpha-hydroxymetoprolol during and after HD

SECONDARY OUTCOMES:
Non-renal clearance phenotype and genotype | Pre-dialysis, during dialysis (30 minutes, 2 hours, end of treatment) and post-dialysis (30 minutes, 2 hours and 4 hours)
  Evaluate the non-renal clearance of metoprolol in patients on HD
Post-dialysis Rebound | post-dialysis (30 minutes, 2 hours and 4 hours)
  Simulate predicted rebound of metoprolol concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Dialysis, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No